CLINICAL TRIAL: NCT01440439
Title: Impact of Insulin Detemir Versus Insulin Glargine on Glycaemic Control and Metabolism During Exercise in Type 1 Diabetes
Brief Title: Comparing Long-acting Insulins During Exercise in Type 1 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buckinghamshire Healthcare NHS Trust (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RXQ425; 2011-001209-28 (EudraCT Number); U1111-1119-8890 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2011-09-20; First posted 2011-09-26 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: insulin glargine; insulin detemir; hypoglycaemia; metabolism; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity | interventions — Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin detemir (Active Comparator): Metabolism during and after submaximal exercise during treatment with insulin detemir
  Interventions: Drug: Insulin detemir
- Insulin glargine (Active Comparator): Metabolism during and after submaximal exercise during treatment with insulin glargine
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin glargine — Use of insulin glargine as basal insulin for treatment of Type 1 Diabetes Mellitus
  Other Names: Lantus
  Arms: Insulin glargine
Drug: Insulin detemir — Use of insulin detemir as basal insulin for treatment of Type 1 Diabetes Mellitus
  Other Names: Levemir
  Arms: Insulin detemir

SUMMARY:
Exercise is an important part of a healthy lifestyle, and many people with Type 1 Diabetes like to take part in regular sport and exercise. The majority of people with Type 1 Diabetes are treated with a "basal bolus" insulin regimen, with background insulin provided by long-acting "basal" insulin doses, and "bolus" doses of short-acting insulin used to accompany food intake. Evidence shows that the main factor preventing people with diabetes from pursuing a more active lifestyle is fear of low blood glucose (hypoglycaemia). A previous study has shown that the type of background insulin affects the likelihood of an individual suffering hypoglycaemia during exercise and for 2 and a half hours afterwards. The aim of this study is to examine this further.

The two most commonly used long-acting insulins, insulin glargine and insulin detemir, will be compared. Previous data suggests that there is a greater likelihood of hypoglycaemia with insulin glargine than insulin detemir. Exercise intensity can have an influence on the likelihood of hypoglycaemia, and in this previous study exercise intensity was measured using heart rate. This study will use a more formal definition of exercise intensity. The investigators will study blood glucose during exercise, but also metabolism as measured by hormones affecting blood glucose levels as well as markers of fat metabolism. The investigators will also use a continuous glucose monitoring system (CGMS) to consider hypoglycaemia on thei night following exercise as this is a recognised consequence of exercise in type 1 diabetes.

The null hypothesis to be tested in this study is that there is no difference between the two insulins in their effect on blood glucose levels and metabolism during exercise and rates of nocturnal hypoglycaemia after exercise.

DETAILED DESCRIPTION:
A1: At the first appointment, potential participants will be screened regarding the inclusion criteria, and if eligible to take part the study information sheet will be discussed with them in detail. Written, informed consent will be obtained if participants are willing to take part in the study. Participants will be given advice and support from this point in order to optimise basal insulin therapy using their usual basal insulin.

A2: Following a period of at least 3 weeks from recruitment into the study, participants will have their maximal oxygen uptake (VO2 MAX - a measure of capacity for physical exercise) assessed.

A3: After at least 4 weeks following recruitment , to allow time for optimisation of basal insulin therapy, and at least one week following A2, the participant's metabolism will then be assessed during and after 60 minutes of exercise at 50% VO2 MAX. Participants will be fitted with a continuous glucose monitoring system (CGMS) to monitor glucose levels for the 24 hours after exercise finishes.

A4: At least 24 hours and no more than 7 days after A3 the participant will switched to using the other trial insulin for basal insulin therapy. Again, participants will be provided with advice and support in order to optimise treatment.

A5: At least 4 weeks following A4, the participant's metabolism will once again be assessed during and after 60 minutes of exercise at 50% VO2 MAX. Participants will again be fitted with CGMS to monitor glucose levels for the 24 hours after exercise finishes.

A6: Once the 24 hours after exercise are complete, the study finishes and participants re-start their usual basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged between 18 and 65 years
* Diagnosed with Type 1 Diabetes Mellitus (T1DM)
* HbA1c < 10% or 86 mmol/mol
* Treated with a basal bolus regimen using either insulin glargine or insulin detemir as the basal insulin
* Exercising regularly for at least 1 hour per week on average

Exclusion Criteria:

* People with any one of the following complications of diabetes:

  * stage 2+ diabetic retinopathy
  * renal impairment (with creatinine >150micromol/l)
  * known history or symptoms of cardiovascular disease
  * foot ulceration
  * peripheral vascular disease
* Pregnancy or breastfeeding
* Untreated or unstable respiratory disease
* Known hypoglycaemia unawareness
* Treatment with drugs known to interfere with glucose metabolism
* Known or suspected allergy to or intolerance of any of the trial drugs or related products
* Receipt of any investigational drug within four months prior to Visit 0
* Known or suspected abuse of alcohol, narcotics or illicit drugs
* Any clinically significant disease or disorder which in the investigator's opinion could interfere with the results of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Glucose excursion (which, as defined below, is the change in blood glucose between the start and finish of one hour of exercise) | Between baseline and 1 hour
  The measure will be a comparison between the two conditions (treatment with insulin detemir or treatment with insulin glargine) of the change in blood glucose levels during one hour of sub-maximal exercise at 50% VO2 MAX

SECONDARY OUTCOMES:
Lactate | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of blood lactate measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
NEFA (Non-esterified fatty acids) | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of NEFA in blood measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
B-OHB (beta-hydroxybutyrate) | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of beta-hydroxybutyrate in blood measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
Catecholamines | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of catecholamines in blood measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
Glucagon | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of glucagon in blood measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
Human growth hormone (hGH) | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of human Growth Hormone in blood measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
Cortisol | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of cortisol in blood measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
IL-6 (interleukin 6) | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of IL-6 in blood measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
High sensitivity CRP (Hs-CRP) | 0, 60 and 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of Hs-CRP in blood measured at the start and the finish of 1 hour of submaximal exercise at 50% VO2 MAX and then 30 minutes following this exercise
RQ (Respiratory Quotient) | Baseline and 1 hour
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of the ratio of RQ measured at the start of exercise to the RQ at the end of 1 hour of submaximal exercise at 50% VO2 MAX
Frequency of hypoglycaemic events | 24 hours
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of the frequency of hypoglycaemic events (defined as blood glucose < 3.5mmol/l) between the start of 1 hour of exercise at 50% VO2 MAX and 24 hours after the end of this exercise.
Time spent in hypoglycaemia | 24 hours
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of the time spent in hypoglycaemia (blood glucose <3.5 mmol/l) between the start of 1 hour of exercise at 50% VO2 MAX and 24 hours after the end of this exercise
Blood glucose | 0, 10, 20, 30, 40, 50, 60, 70, 80, 90 minutes
  This measure consists of a comparison between the two conditions (treatment with insulin glargine and treatment with insulin detemir) of blood glucose levels measured every 10 minutes from the start of 1 hour of submaximal exercise at 50% VO2 MAX until 30 minutes following this exercise

CONTACTS AND LOCATIONS:
Overall Officials: Ian W Gallen, MD FRCP, Principal Investigator — Bcukinghamshire Healthcare NHS Trust
Locations (1):
- Wycombe Hospital, High Wycombe, Buckinghamshire, United Kingdom